CLINICAL TRIAL: NCT00974064
Title: The Natural History of Gene Expression in Lung Cells of Non-Smokers, Smokers, and Ex-Smokers in Health and Disease
Brief Title: The Natural History of Gene Expression in the Lung Cells of Non-Smokers, Smokers and Ex-Smokers in Health and Disease
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 0905010391
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Smoking; Smoking Cessation; Chronic Bronchitis; Emphysema
Keywords: COPD; Lung disease; Chronic bronchitis; Emphysema; Smoking; Smoking cessation; Quit smoking; Healthy smoker; Smoker; Non-smoker
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Smoking; Smoking Cessation; Bronchitis, Chronic; Emphysema; Lung Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Subjects will not have more than 550 mL of blood drawn over a period of 8 weeks. Airway epithelium from airway brushing samples and alveolar macrophages from bronchoalveolar lavage is processed to yield high quality RNA. Complimentary DNA (cDNA) is transcribed from the RNA in vitro and the product is hybridized onto gene microarray chips.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- A-Healthy Non smokers: Healthy nonsmokers. Defined as non-smokers by self report and urine cotinine levels consistent with a nonsmoker (urine cotinine <5 ng/mL).
- B-Healthy smoker: Healthy current smokers. Subjects categorized as healthy according to criteria under "Collection" (#1204012331) protocol.
- C-Healthy smoker to quit: Healthy smokers willing to quit. Defined by self-report and urine cotinine levels consistent with an active smoker (urine cotinine >50 ng/mL).
- D-Current smoker w. COPD: Current smokers with COPD. COPD as defined by the GOLD criteria and currently smoking as defined by self-report and urine cotinine levels consistent with an active smoker (urine cotinine >50 ng/mL)
- E-Current COPD smoker to quit: Current smokers with COPD willing to stop smoking. Subjects have COPD as defined by the GOLD criteria

SUMMARY:
Cigarette smoking is the major risk factor for chronic obstructive pulmonary disease (COPD, commonly known as chronic bronchitis and emphysema). Despite this clear link, only 15-20% of smokers develop COPD suggesting that genetic factors affect the lung's susceptibility to the stress of cigarette smoke. The cells lining the airways (epithelium) and cells that help defend the lung (alveolar macrophages) of smokers develop gene expression changes that are different from that of nonsmokers. In the investigators' previous studies they have demonstrated that there are greater than 200 genes that are responsive to cigarette smoke in these cells. But the investigators do not know whether the gene expression is static or changes as a function of time. Genes that show significant changes over time may be relevant to the progression of the disease. Even though quitting smoking reduces the rate at which the lungs decline, many-smokers still go on to develop COPD. This study will provide insights into the natural history of smoking-related gene expression of the lung cells in health and disease.

DETAILED DESCRIPTION:
Cigarette smoke is responsible for the majority of lung cancers and is the major cause of COPD, the fourth leading cause of death in the United States. Despite the well established causal role of cigarette smoking in lung cancer and COPD, only 10-20% of smokers actually develop these diseases. This suggests that there are genetic predisposing factors that place some individuals at greater risk. Our prior work shows that healthy smokers (cigarette smokers with normal history, physical exam, lung function tests and chest x-rays) and smokers with COPD have marked up and down regulation of greater than 200 genes in the small airway epithelium and alveolar macrophages. There is however, a varied response to smoking among individuals, with some individuals abnormally expressing far fewer genes. The focus of this study is to evaluate the hypothesis that the response of the lung cells to the stress of smoking is unique to each individual but is consistent over time. Furthermore, individuals that stop smoking will each have a unique response, but is constant over time for each individual. By defining the patterns of biologic response over time among smoking, ex-smoking and nonsmoking subjects, we will be able to identify common biologic pathways as potential targets for intervention.

ELIGIBILITY:
Inclusion Criteria:

Group A: Healthy nonsmokers

* All study individuals should be enrolled in the "Airway" protocol #1204012331 "Collection of Airway, Blood and/or Urine Specimens from Subjects for Research Studies"
* Willing and able to provide informed consent for the long term follow up study with repeated bronchoscopies
* Male and Female subject ≥18 years of age
* Never smokers is defined as someone who has smoked < 100 cigarettes per lifetime and whose urine nicotine <2 ng/mL and/or urine cotinine <5 ng/mL, at entry into the study

Group B: Healthy current smokers Inclusion:

* All study individuals should be enrolled in the "Airway" protocol
* Willing and able to provide informed consent for the long term follow up study with repeated bronchoscopies
* Male and Female subject ≥18 years of age
* Active smoker as evidenced by self-report and urine nicotine >30 ng/mL and/or urine cotinine >50 ng/mL

Group C: Healthy smokers who elect to stop smoking Inclusion:

* All study individuals should be enrolled in the "Airway" protocol
* Willing and able to provide informed consent for the long term follow up study with repeated bronchoscopies
* Male and Female subject ≥18 years of age
* Current smoker as evidenced by self-report and urine nicotine >30 ng/mL and/or urine cotinine >50 ng/mL
* Be a current smoker willing to stop smoking

Group D - Current smokers with COPD Inclusion:

* All study subjects will be enrolled in the "Airway" protocol #1204012331 "Collection of Airway, Blood and/or Urine Specimens from Subjects for Research Studies"
* All study subjects should meet the lung disease criteria for having COPD may be of any stage (GOLD I - IV), be ambulatory and have no evidence of respiratory failure
* All study subjects should be able to provide informed consent for the long term follow up study with repeated bronchoscopies
* Male and Female subject ≥18 years of age
* Active smokers as evidenced by urine nicotine >30 ng/mL and/or urine cotinine >50 ng/mL

Group E - Current smokers with COPD who elect to stop smoking Inclusion:

* All study subjects will be enrolled in the "Airway" protocol #1204012331 "Collection of Airway, Blood and/or Urine Specimens from Subjects for Research Studies"
* All study subjects should meet the lung disease criteria for having COPD may be of any stage (GOLD I - IV), be ambulatory and have no evidence of respiratory failure
* All study subjects should be able to provide informed consent for the long term follow up study with repeated bronchoscopies
* Male and Female subject ≥18 years of age
* Active smokers as evidenced by urine nicotine >30 ng/mL and/or urine cotinine >50 ng/mL
* Be a current smoker willing to stop smoking

Exclusion Criteria:

Groups A - E

* Individuals unable to provide proper informed consent
* Habitual use of drugs and/or alcohol within the past six months (Acceptable: Marijuana one time in three months; average of two alcoholic beverages per day; drug and/or alcohol abuse is defined as per the DSM-IV Substance Abuse Criteria)
* Individuals with asthma and with recurrent or recent (within three months) and/or acute pulmonary infection
* Individuals with allergy to lidocaine
* Significant kidney disease or subjects on dialysis
* Females who are pregnant or lactating or intending to become pregnant in the next 12 months
* Subjects who are HIV positive
* Subjects that have unstable coronary artery disease as evidenced by unstable angina, >Class II New York Heart Association (NYHA) cardiac status, history of congestive heart failure or MI within the last 12 months
* Subjects who are contraindicated for undergoing bronchoscopy
* Subjects having any medical condition that in the opinion of the investigator would preclude the subject from entering the study

Groups D and E

- Subjects may not have evidence of respiratory failure such as SpO2 <90% or PaO2 <60 mmHg

Groups C and E

* Current major depression or other significant psychiatric disorder
* Subjects currently taking anti-depressant medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: New York Metropolitan area residents
Sampling Method: Non-Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Evaluate gene expression over time | 12/31/2013
  To prospectively assess changes in lung cell gene expression over time in healthy nonsmokers, healthy smokers and smokers with COPD. To examine what smoking-induced gene expression changes occur in the lung cells of healthy smokers and COPD smokers over time in response to cessation of smoking.

SECONDARY OUTCOMES:
Quitters who return to smoking and the effects on gene expression | 12/31/2012
  In individuals who quit but start smoking again despite the standard smoking cessation therapy, what are the effects on gene expression of returning to smoking. To assess whether baseline gene expression determines what genes rapidly change to a more "normal" expression pattern with smoking cessation. Does having established COPD determine the relative reversibility of the gene expression pattern with smoking cessation compared to healthy smokers.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G. Crystal, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College and Weill Cornell Medical Center, Department of Genetic Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Strulovici-Barel Y, Staudt MR, Krause A, Gordon C, Tilley AE, Harvey BG, Kaner RJ, Hollmann C, Mezey JG, Bitter H, Pillai SG, Hilton H, Wolff G, Stevenson CS, Visvanathan S, Fine JS, Crystal RG. Persistence of circulating endothelial microparticles in COPD despite smoking cessation. Thorax. 2016 Dec;71(12):1137-1144. doi: 10.1136/thoraxjnl-2015-208274. Epub 2016 Jul 26. PMID 27462120